CLINICAL TRIAL: NCT04756622
Title: Efficacy and Safety of N-acetyl Cysteine for the Prevention of Oral Mucositis After High-dose Chemotherapy and Autologous Hematopoietic Cell Transplantation: a Phase III, Randomized, Open Label, Multi-center Study.
Brief Title: N-acetyl Cysteine for the Prevention of Oral Mucositis After Autologous Hematopoietic Cell Transplantation.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: moshe yeshurun (Other)
Responsible Party: Sponsor-Investigator, moshe yeshurun, Head Bone Marrow UNit, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1078-20
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Mucositis; Transplant-Related Disorder
MeSH Terms: conditions — Mucositis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Phase III, randomized, open label and multi-center study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N acetyl cysteine (Experimental): NAC dissolved in water at a dose of 600 mg three times per day from day of transplant until neutrophil engraftment, or upon resolution of OM, whichever appears later.
  Interventions: Drug: N acetyl cysteine
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: N acetyl cysteine — N acetyl cysteine dissolved in water at a dose of 600 mg three times daily from day of transplant until neutrophil engraftment, or upon resolution of OM, whichever appears later.
  Arms: N acetyl cysteine

SUMMARY:
Oral mucositis (OM) is a major source of morbidity in patients undergoing hematopoietic cell transplantation (HCT). N-acetyl cysteine (NAC) is an antioxidant, widely used as mucolytic agent or antidote of acetaminophen overdose hepatotoxicity. we intend to explore the safety and efficacy of NAC in the prevention of OM after high-dose chemotherapy and autologous HCT in a phase III, randomized, open label and multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma and lymphoma in partial response and complete remission.
* Undergoing high-dose chemotherapy with autologous transplantation.

Exclusion Criteria:

• Known sensitivity to NAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with grade 3-4 OM | day 14
  Proportion of patients with grade 3-4 OM

SECONDARY OUTCOMES:
Proportion of patients with grade 1-4 OM | 14 days
  Proportion of patients with grade 1-4 OM
Time from transplantation to first hospital discharge | 30 days
  Time from transplantation to first hospital discharge
Non-relapse mortality | day 50
  Non-relapse mortality

IPD SHARING:
Plan to Share IPD: No